CLINICAL TRIAL: NCT00252018
Title: The Effect of Broccoli Sprouts as a Nutritional Supplement in the Prevention of Cardiovascular Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KF 01-257/04
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus; Hypertension; Hypercholesterolemia; Cardiovascular Disease
Keywords: Nutritional supplement; Prevention; Endothelial function; Flow mediated dilation
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hypercholesterolemia; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Daily intake of broccoli sprouts

SUMMARY:
The purpose of this study is to investigate whether a daily intake of dried broccoli sprouts will improve the endothelial function of the participants as measured by Flow mediated dilation (FMD)

The dried sprouts are chosen because broccoli sprouts are known as containing large amounts af the glucosinolate glucoraphanin which in vitro and in animal models has been shown to have a positive effect on the endothelium as measured by NO release.

DETAILED DESCRIPTION:
Inflammation plays an important role in the development of atherosclerosis. The initial site of damage is the endothelium and secondarily the rest of the vascular wall is involved. Hypotheses concerning the development of these lesions have introduced the concept of oxidative stress, ("an imbalance between oxidants and antioxidants in favor of the oxidants, potentially leading to damage") as having a key role in the development of atherosclerosis. Consequently, much interest has been focused on attenuating oxidative stress in order to minimize this damage.

Clinical trials for the study of the effect of antioxidants on the atherosclerotic process, using micronutrients with a reductive potential, have failed to demonstrate a benefit for the patients and some have even shown an increased mortality.

An alternative is to induce the endogenous antioxidative defense of the cell. One possibility is to increase the expression of enzymes responsible for neutralizing oxidative substances, a group of enzymes relevant for this path are the phase 2 enzymes, for instance gluthation-s-transferase(GsT).

Broccoli sprouts have a very high content of Glucoraphanin(GP) a substance which has the ability to increase the expression of GsT.

Experiments involving stroke prone hypertensive rats and humans have indicated that GP in broccoli sprouts have a beneficial effect against oxidative stress. In the experiment with the rats a consequence of the protection against oxidative stress was an increase in endothelial dependant vasodilation(EDV). This finding is important because low EDV predicts development of atherosclerosis.

We find that induction of enzymes with antioxidant capabilities could be beneficial for people with atherosclerosis and that a study of the effects of broccoli sprouts on endothelial function in conditions with endothelial dysfunction are important as an intermediary step before clinical studies are performed.

Hypothesis Broccoli sprouts containing high levels of GP induce phase 2 enzymes in the human endothelium, thereby making the endothelium more resistant to inflammatory damage. Attenuation of damage should increase nitric oxide (NO) bioavailability and thus improve EDV of patients being in risk of cardiovascular disease.

Methods Broccoli sprouts will be harvested after 4 days to obtain the highest amount of GP per unit of dry weight. After harvesting, the sprouts will be dried in order to avoid degradation of the GP content. As placebo, sprouts where the GP content is degraded will be used.

The participants will receive 10 g dried broccoli sprouts per day for a period of four weeks. 10 g dried sprouts has a GP content equivalent to the content of 1 to 10 kg of fresh broccoli.

Blinding of the participants as well as the investigators will be insured.

Participants:

120 patients in three subgroups and 40 healthy controls giving a total of four groups.

The groups will be investigated individually, having each a treatment and a placebo arm.

Patients will be screened during which interview BP, weight height and blood test will be performed. After informed consent is obtained, they will be randomized by draw of an envelope to either placebo or active ingredient. At the beginning of the study and every other week during the study, the patients will be examined by BP, weight, blood samples and assessment of EDV by use of flow mediated dilation(FMD).

FMD will be performed by measuring increase of diameter of the brachial artery above the elbow before and after interruption of circulation to the forearm for a period of 5 minutes by use of a tourniquet placed below the elbow. Flow through the brachial artery will be recorded immediately after circulation is restored for 15 s. Dilation will be expressed as a ratio relative to the diameter prior to interruption in percent. Blood samples will be analyzed for GP content and metabolites at KVL.

Statistics We have determined σ in our studies to be less than 2.5 which is comparable to results form other groups. Assuming a σ of 3 and a minimal detectable difference of 3% (usually the FMD is approximately 5%) will give a power of >85% when the level of significance is 5% with our group size.

Ethics WE find the participants will have no risks and only minor inconveniences when participating in our study.

The study is approved by the Ethics committee of Copenhagen and Frederiksberg Municipalities (no 01-257/04).

The study will be published in a peer reviewed biomedical journal

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from hypertension, having a diastolic blood pressure of above 90 mm Hg or a systolic blood pressure of more than 140 mm Hg.
* Patients suffering from NIDDM, according to present criteria for diagnosis of NIDDM:
* People with dyslipidemia (combination of total cholesterol above 5, LDL cholesterol above 3 and HDL cholesterol below 1.1)
* Healthy controls suffering from none of the above conditions, but otherwise (age, sex, BMI and lifestyle) corresponding to the patient groups.

Exclusion Criteria:

* Patients under the age of 18 at inclusion in the study.
* Pregnant or breastfeeding women
* Women of childbearing age with no safe method of contraception
* Patients receiving vitamin K-antagonists (coumarine, marcoumar etc)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Improvement of endothelial function as measured by FMD

CONTACTS AND LOCATIONS:
Overall Officials: Christian Torp-Pedersen, MD, Study Chair — Bispebjerg Hospital Department of Cardiology
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Wu L, Noyan Ashraf MH, Facci M, Wang R, Paterson PG, Ferrie A, Juurlink BH. Dietary approach to attenuate oxidative stress, hypertension, and inflammation in the cardiovascular system. Proc Natl Acad Sci U S A. 2004 May 4;101(18):7094-9. doi: 10.1073/pnas.0402004101. Epub 2004 Apr 21. PMID 15103025
- [Background] Murashima M, Watanabe S, Zhuo XG, Uehara M, Kurashige A. Phase 1 study of multiple biomarkers for metabolism and oxidative stress after one-week intake of broccoli sprouts. Biofactors. 2004;22(1-4):271-5. doi: 10.1002/biof.5520220154. PMID 15630296
- [Background] Fahey JW, Zhang Y, Talalay P. Broccoli sprouts: an exceptionally rich source of inducers of enzymes that protect against chemical carcinogens. Proc Natl Acad Sci U S A. 1997 Sep 16;94(19):10367-72. doi: 10.1073/pnas.94.19.10367. PMID 9294217
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Brunner H, Cockcroft JR, Deanfield J, Donald A, Ferrannini E, Halcox J, Kiowski W, Luscher TF, Mancia G, Natali A, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Spieker LE, Taddei S, Webb DJ; Working Group on Endothelins and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part II: Association with cardiovascular risk factors and diseases. A statement by the Working Group on Endothelins and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Feb;23(2):233-46. doi: 10.1097/00004872-200502000-00001. PMID 15662207
- [Background] Matusheski NV, Juvik JA, Jeffery EH. Heating decreases epithiospecifier protein activity and increases sulforaphane formation in broccoli. Phytochemistry. 2004 May;65(9):1273-81. doi: 10.1016/j.phytochem.2004.04.013. PMID 15184012
- [Background] Stocker R, Keaney JF Jr. Role of oxidative modifications in atherosclerosis. Physiol Rev. 2004 Oct;84(4):1381-478. doi: 10.1152/physrev.00047.2003. PMID 15383655
- [Derived] Christiansen B, Bellostas Muguerza N, Petersen AM, Kveiborg B, Madsen CR, Thomas H, Ihlemann N, Sorensen JC, Kober L, Sorensen H, Torp-Pedersen C, Dominguez H. Ingestion of broccoli sprouts does not improve endothelial function in humans with hypertension. PLoS One. 2010 Aug 27;5(8):e12461. doi: 10.1371/journal.pone.0012461. PMID 20805984